CLINICAL TRIAL: NCT02988401
Title: Intranasal Insulin for Improving Cognitive Function in Multiple Sclerosis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00095554
Record Dates: First submitted 2016-12-07; First posted 2016-12-09 (Estimated); Results first posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-02

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Secondary Progressive; Multiple Sclerosis, Primary Progressive
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Intranasal insulin 20 international units (Experimental): Subjects will administer 20 I.U. of insulin in the nostrils using a ViaNaseTM controlled particle dispersion nasal device two times/day (BID) for 24 weeks.
  Interventions: Drug: Insulin
- Intranasal insulin 10 international units (Experimental): Subjects will administer 10 I.U. of insulin in the nostrils using a ViaNaseTM controlled particle dispersion nasal device two times/day (BID) for 24 weeks.
  Interventions: Drug: Insulin
- Intranasal saline (Placebo Comparator): Subjects will administer a sterile diluent containing inactive ingredients in the nostrils using a ViaNaseTM controlled particle dispersion nasal device two times/day (BID) for 24 weeks.
  Interventions: Drug: Placebo (Sterile diluent)

INTERVENTIONS:
Drug: Insulin — All patients will receive either insulin or placebo using the Vianase III N2B device during the first 24 weeks of the study.
  Arms: Intranasal insulin 10 international units; Intranasal insulin 20 international units
Drug: Placebo (Sterile diluent) — All patients will receive either insulin or placebo using Vianase III N2B device during the first 24 weeks of the study.
  Arms: Intranasal saline

SUMMARY:
This study will evaluate if giving insulin that is administered in the nostrils (intranasal) is safe and tolerable for people with multiple sclerosis (MS). It is also being done to evaluate if intranasal insulin improves cognitive function in people with MS and to evaluate how it might be working.

DETAILED DESCRIPTION:
Cognitive impairment is common in and devastating to people with MS. MS is a common, chronic, central nervous system (CNS) disease characterized by inflammation, demyelination, and neurodegeneration. One of the most devastating symptoms of this disease is impaired cognitive function, which is common and present in over 60% of individuals with MS. MS-related cognitive impairment is associated with lowered quality of life and reduced functional capacity, including loss of employment, impaired social relationships, compromised driving safety, and poor adherence to treatment. Impaired cognitive functioning has been observed early in the disease, sometimes even before diagnosis, and cognitive function has been shown to decline longitudinally, both over the short- and long-term. Several cognitive domains are impacted in people with MS, including attention, memory, executive functioning, and especially processing speed.

To date, multiple pharmacologic interventions have been assessed with disappointing results. There was no significant difference between treatment and placebo for cognition in randomized control trials of donepezil, aminopyridines, gingko biloba, and memantine. Psychostimulants demonstrated some efficacy, but only in secondary outcome measures. Behavioral interventions show promise but are understudied. Furthermore, cognitive rehabilitation is often time consuming, costly, and not universally available. Hence, there is an urgent need to identify or develop novel therapies that can help improve cognitive function in MS.

Intranasal insulin is extremely safe and tolerable in other populations, allowing for concentrated delivery to the nervous system. An intranasal delivery system provides a non-invasive way to bypass the blood-brain barrier and allow rapid delivery of a medication to the CNS via the olfactory and trigeminal perivascular channels.The main advantage of the delivery system is reducing systemic side effects via limiting a medication's exposure to peripheral organs and tissues.

Insulin administration has been shown to improve memory and learning in healthy people and in those with neurodegenerative diseases. Intranasal insulin has been shown to have neuroprotective and restorative effects in several human clinical trials. Overall, findings suggest that intranasal insulin not only affects cognitive function acutely, but that over time, there may be associated structural changes that lead to a more permanent treatment benefit. Cognitive dysfunction is very common in MS and can be devastating, therefore a treatment intervention (i.e., intranasal insulin) can help both acutely and longitudinally.

The primary aim of this study is to assess the safety and tolerability of intranasal insulin in people with MS. The secondary aim is to evaluate if intranasal insulin improves learning and memory in people with MS. The third aim is to evaluate the impact of intranasal insulin on measures of oxidative stress, axonal injury, cellular stress, and energy metabolism in MS.

ELIGIBILITY:
Inclusion Criteria:

* Meets 2010 criteria for MS
* No relapse in past 3 months
* At least mild cognitive impairment (based off of SDMT/PST score)
* Capacity to learn and self-administer intranasal insulin/placebo, or presence of a caregiver with such capacity who is willing to do it for the duration of the trial
* Untreated/on the same MS therapy for at least 6 months, with no anticipated change in the next year
* Willing to prevent pregnancy during study if female of childbearing potential

Exclusion Criteria:

* Current, active major depression
* No tricyclic antidepressant or anticonvulsant (except carbamazepine, pregabalin or gabapentin) use within 6 weeks of screening; if on oxybutynin or tolterodine, on stable dose for > 6 months without plans for changing dose in next year
* If taking selective serotonin (± norepinephrine) reuptake inhibitors, pregabalin, gabapentin, sympathomimetic, monoamine oxidase inhibitor, antipsychotic, amantadine, cholinesterase inhibitor, memantine, modafanil, armodafinil, or evening short-acting benzodiazepines, on stable dose for 6 weeks or greater
* Pregnant or nursing
* THC; illicit drug or alcohol abuse in past 3 months
* History of diabetes mellitus or insulin resistance
* Active liver disease, stage IV/V kidney disease or severe metabolic derangements
* CNS disorder other than MS or headache

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mowry, MD, MCR, Principal Investigator — Johns Hopkins University; Scott Newsome, DO, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benedict RH, Cookfair D, Gavett R, Gunther M, Munschauer F, Garg N, Weinstock-Guttman B. Validity of the minimal assessment of cognitive function in multiple sclerosis (MACFIMS). J Int Neuropsychol Soc. 2006 Jul;12(4):549-58. doi: 10.1017/s1355617706060723. PMID 16981607
- [Background] DeLuca J. What we know about cognitive changes in multiple sclerosis. In: LaRocca N, Kalb R, eds. Multiple Sclerosis: Understanding the Cognitive Challenges. New York: Demos Health; 2006: 17-40.
- [Background] Rao S. Cognitive Function in Patients with Multiple Sclerosis: Impairment and Treatment. IJMSC 2004;1:9-22.
- [Background] Ruet A, Deloire M, Hamel D, Ouallet JC, Petry K, Brochet B. Cognitive impairment, health-related quality of life and vocational status at early stages of multiple sclerosis: a 7-year longitudinal study. J Neurol. 2013 Mar;260(3):776-84. doi: 10.1007/s00415-012-6705-1. Epub 2012 Oct 19. PMID 23081755
- [Background] Strober LB, Christodoulou C, Benedict RH, Westervelt HJ, Melville P, Scherl WF, Weinstock-Guttman B, Rizvi S, Goodman AD, Krupp LB. Unemployment in multiple sclerosis: the contribution of personality and disease. Mult Scler. 2012 May;18(5):647-53. doi: 10.1177/1352458511426735. Epub 2011 Dec 19. PMID 22183935
- [Background] Morrow SA, Drake A, Zivadinov R, Munschauer F, Weinstock-Guttman B, Benedict RH. Predicting loss of employment over three years in multiple sclerosis: clinically meaningful cognitive decline. Clin Neuropsychol. 2010 Oct;24(7):1131-45. doi: 10.1080/13854046.2010.511272. Epub 2010 Sep 8. PMID 20830649
- [Background] Schultheis MT, Weisser V, Ang J, Elovic E, Nead R, Sestito N, Fleksher C, Millis SR. Examining the relationship between cognition and driving performance in multiple sclerosis. Arch Phys Med Rehabil. 2010 Mar;91(3):465-73. doi: 10.1016/j.apmr.2009.09.026. PMID 20298841
- [Background] Patti F. Optimizing the benefit of multiple sclerosis therapy: the importance of treatment adherence. Patient Prefer Adherence. 2010 Feb 4;4:1-9. doi: 10.2147/ppa.s8230. PMID 20165593
- [Background] Rao SM, Leo GJ, Ellington L, Nauertz T, Bernardin L, Unverzagt F. Cognitive dysfunction in multiple sclerosis. II. Impact on employment and social functioning. Neurology. 1991 May;41(5):692-6. doi: 10.1212/wnl.41.5.692. PMID 1823781
- [Background] Amato MP, Razzolini L, Goretti B, Stromillo ML, Rossi F, Giorgio A, Hakiki B, Giannini M, Pasto L, Portaccio E, De Stefano N. Cognitive reserve and cortical atrophy in multiple sclerosis: a longitudinal study. Neurology. 2013 May 7;80(19):1728-33. doi: 10.1212/WNL.0b013e3182918c6f. Epub 2013 Apr 10. PMID 23576622
- [Background] Amato MP, Ponziani G, Siracusa G, Sorbi S. Cognitive dysfunction in early-onset multiple sclerosis: a reappraisal after 10 years. Arch Neurol. 2001 Oct;58(10):1602-6. doi: 10.1001/archneur.58.10.1602. PMID 11594918
- [Background] Lacy M, Hauser M, Pliskin N, Assuras S, Valentine MO, Reder A. The effects of long-term interferon-beta-1b treatment on cognitive functioning in multiple sclerosis: a 16-year longitudinal study. Mult Scler. 2013 Nov;19(13):1765-72. doi: 10.1177/1352458513485981. Epub 2013 May 7. PMID 23652214
- [Background] DeLuca J, Barbieri-Berger S, Johnson SK. The nature of memory impairments in multiple sclerosis: acquisition versus retrieval. J Clin Exp Neuropsychol. 1994 Apr;16(2):183-9. doi: 10.1080/01688639408402629. PMID 8021305
- [Background] DeLuca J, Gaudino EA, Diamond BJ, Christodoulou C, Engel RA. Acquisition and storage deficits in multiple sclerosis. J Clin Exp Neuropsychol. 1998 Jun;20(3):376-90. doi: 10.1076/jcen.20.3.376.819. PMID 9845164
- [Background] Thornton AE, Raz N, Tucke KA. Memory in multiple sclerosis: contextual encoding deficits. J Int Neuropsychol Soc. 2002 Mar;8(3):395-409. doi: 10.1017/s1355617702813200. PMID 11939698
- [Background] DeLuca J, Chelune GJ, Tulsky DS, Lengenfelder J, Chiaravalloti ND. Is speed of processing or working memory the primary information processing deficit in multiple sclerosis? J Clin Exp Neuropsychol. 2004 Jun;26(4):550-62. doi: 10.1080/13803390490496641. PMID 15512942
- [Background] Demaree HA, DeLuca J, Gaudino EA, Diamond BJ. Speed of information processing as a key deficit in multiple sclerosis: implications for rehabilitation. J Neurol Neurosurg Psychiatry. 1999 Nov;67(5):661-3. doi: 10.1136/jnnp.67.5.661. PMID 10519876
- [Background] Krupp LB, Christodoulou C, Melville P, Scherl WF, Pai LY, Muenz LR, He D, Benedict RH, Goodman A, Rizvi S, Schwid SR, Weinstock-Guttman B, Westervelt HJ, Wishart H. Multicenter randomized clinical trial of donepezil for memory impairment in multiple sclerosis. Neurology. 2011 Apr 26;76(17):1500-7. doi: 10.1212/WNL.0b013e318218107a. PMID 21519001
- [Background] Solari A, Uitdehaag B, Giuliani G, Pucci E, Taus C. Aminopyridines for symptomatic treatment in multiple sclerosis. Cochrane Database Syst Rev. 2001;2002(4):CD001330. doi: 10.1002/14651858.CD001330. PMID 11687106
- [Background] Lovera JF, Kim E, Heriza E, Fitzpatrick M, Hunziker J, Turner AP, Adams J, Stover T, Sangeorzan A, Sloan A, Howieson D, Wild K, Haselkorn J, Bourdette D. Ginkgo biloba does not improve cognitive function in MS: a randomized placebo-controlled trial. Neurology. 2012 Sep 18;79(12):1278-84. doi: 10.1212/WNL.0b013e31826aac60. Epub 2012 Sep 5. PMID 22955125
- [Background] Lovera JF, Frohman E, Brown TR, Bandari D, Nguyen L, Yadav V, Stuve O, Karman J, Bogardus K, Heimburger G, Cua L, Remingon G, Fowler J, Monahan T, Kilcup S, Courtney Y, McAleenan J, Butler K, Wild K, Whitham R, Bourdette D. Memantine for cognitive impairment in multiple sclerosis: a randomized placebo-controlled trial. Mult Scler. 2010 Jun;16(6):715-23. doi: 10.1177/1352458510367662. Epub 2010 May 18. PMID 20483885
- [Background] Morrow SA, Kaushik T, Zarevics P, Erlanger D, Bear MF, Munschauer FE, Benedict RH. The effects of L-amphetamine sulfate on cognition in MS patients: results of a randomized controlled trial. J Neurol. 2009 Jul;256(7):1095-102. doi: 10.1007/s00415-009-5074-x. Epub 2009 Mar 5. PMID 19263186
- [Background] Mitolo M, Venneri A, Wilkinson ID, Sharrack B. Cognitive rehabilitation in multiple sclerosis: A systematic review. J Neurol Sci. 2015 Jul 15;354(1-2):1-9. doi: 10.1016/j.jns.2015.05.004. Epub 2015 May 9. PMID 25998261
- [Background] Craft S, Baker LD, Montine TJ, Minoshima S, Watson GS, Claxton A, Arbuckle M, Callaghan M, Tsai E, Plymate SR, Green PS, Leverenz J, Cross D, Gerton B. Intranasal insulin therapy for Alzheimer disease and amnestic mild cognitive impairment: a pilot clinical trial. Arch Neurol. 2012 Jan;69(1):29-38. doi: 10.1001/archneurol.2011.233. Epub 2011 Sep 12. PMID 21911655

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Subjects will administer a sterile diluent containing inactive ingredients in the nostrils using a ViaNaseTM controlled particle dispersion nasal device two times/day (BID) for 24 weeks.
  Placebo (Sterile diluent): All patients will receive either insulin or placebo using Vianase III N2B device during the first 24 weeks of the study.
Period: Overall Study
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Started | 37 | 33 | 35
Completed (There were 69 total participants that had at least one follow-up visit up until week 24.) | 24 | 17 | 28
Not Completed | 13 | 16 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo | Total
Number analyzed (Participants) | 37 | 33 | 35 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.5 (10.1) | 54.4 (9.2) | 49.4 (9.2) | 52.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 22 | 65
  Male | 17 | 10 | 13 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 8 | 11 | 31
  White | 25 | 25 | 24 | 74
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 37 | 33 | 35 | 105

OUTCOME MEASURES:

1. Primary Outcome: Change in Cognitive Function as Assessed by the Symbol Digit Modalities Test (SDMT)
Description: This task will be performed at five study visits. The SDMT is one of the most commonly used tests to assess processing speed in the MS population and is included in the Minimal Assessment of Cognitive Function in MS (MACFIMS). Higher scores reflect a better outcome (range 0 to 110). In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the primary analyses include the SDMTs acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the SDMT.
Time Frame: Up to week 24 visit
Population: Individuals with pre-treatment SDMT were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 32 | 30 | 32
score on a scale | 0.145 [0.000 to 0.290] | 0.207 [0.033 to 0.381] | 0.163 [0.029 to 0.297]

2. Secondary Outcome: Number of Participants With Adverse Events Leading to Study Discontinuation
Description: An adverse event will be defined as any occurrence or worsening of an undesirable or unintended sign, symptom (or abnormal laboratory test), or disease temporally associated with the use of a medicinal product or intervention, whether or not it is considered related to the product/intervention. We report overall adverse events in the relevant section. Here, we report adverse events that led to study discontinuation.
Time Frame: Up to week 24 visit
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 37 | 33 | 35
Participants | 3 | 2 | 1

3. Secondary Outcome: Fingerstick Blood Glucose (Subset)
Description: Fingerstick blood glucose levels were monitored twice within the 90 minutes following the first dose administration of study drug for the first 15 participants.
Time Frame: At the baseline visit, monitored twice within the 90 minutes following the first dose administration of study drug
Population: The first 15 participants were included in this safety substudy. One placebo participant was missing the second measurement.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 5 | 5 | 5
mg/dL
  First timepoint | 97.8 (13.4) | 95.8 (15.5) | 90.0 (18.4)
  Second timepoint: number analyzed (Participants) | 5 | 5 | 4
  Second timepoint | 88.4 (8.8) | 92.2 (15.5) | 87.8 (11.4)

4. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Controlled Oral Word Association Test (COWAT)
Description: This test measures phonemic fluency. The test scores the number of words a participant can provide that begin with a specified letter within one minute, such that scores range from zero (worst) to an infinite number (better). Total score is sum of three 60-second trials. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the primary analyses include the COWAT scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 37 | 31 | 35
score on a scale | 0.090 [-0.112 to 0.292] | 0.070 [-0.162 to 0.303] | 0.021 [-0.174 to 0.216]

5. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the California Verbal Learning Test, Second Edition (CVLT-II)
Description: This is a verbal learning and memory test. Scores range from zero to 16; a higher number is better. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the primary analyses include the CVLT-II scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 36 | 31 | 35
score on a scale | 0.082 [0.015 to 0.149] | 0.021 [-0.057 to 0.100] | 0.020 [-0.043 to 0.082]

6. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Brief Visuospatial Memory Test - Revised (BVMT-R) Delayed Recall
Description: This is a visual, nonverbal test of learning and memory. Scores range from zero to 12; higher is better. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include the BVMT-R delayed recall scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 36 | 29 | 34
score on a scale | 0.027 [-0.020 to 0.074] | 0.059 [0.006 to 0.113] | 0.030 [-0.015 to 0.075]

7. Secondary Outcome: Change in Cognitive Function as Assessed by the Rao-version of the Paced Auditory Serial Addition Test (PASAT)
Description: The Rao-version of the PASAT evaluates processing speed, working memory, and basic addition skills. Scores range from zero to 60; higher is better. Herein we present 3-second PASAT results ("PASAT-3"). In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include PASAT-3 scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the SDMT.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 36 | 29 | 30
score on a scale | 0.372 [0.180 to 0.563] | 0.363 [0.136 to 0.591] | 0.212 [0.027 to 0.398]

8. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Judgement of Line Orientation Test (JLO)
Description: Judgment of Line Orientation Test measures a person's ability to match the angle and orientation of lines in space. Scores range from zero to 30; higher is better. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include JLO data acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 36 | 29 | 35
score on a scale | -0.031 [-0.109 to 0.046] | 0.047 [-0.044 to 0.139] | -0.005 [-0.079 to 0.069]

9. Secondary Outcome: Change From Baseline in Cognitive Function as Assessed by the Delis-Kaplan Executive Function System Sorting Test
Description: This test measures executive functioning, concept formation, and cognitive flexibility. Scores range from zero to 16; higher is better. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include DKEFS correct sort scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline assessment were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 35 | 29 | 32
score on a scale | -0.001 [-0.112 to 0.111] | 0.027 [-0.104 to 0.159] | 0.002 [-0.114 to 0.118]

10. Other Pre Specified Outcome: Assess Depression Severity, as Measured by the Beck Depression Inventory-II (BDI-II)
Description: The BDI-II is a 21-question multiple-choice self-report inventory test for measuring the severity of depression. Scores range from zero to 63; higher scores indicate greater depression. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include the BDI-II scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the scores.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline questionnaire were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 31 | 25 | 27
score on a scale | -0.022 [-0.152 to 0.108] | -0.019 [-0.179 to 0.140] | -0.045 [-0.183 to 0.094]

11. Other Pre Specified Outcome: Evaluation of Impact of Study Products on Health Related Quality of Life Using the Functional Assessment of Multiple Sclerosis Questionnaire (FAMS)
Description: FAMS is a self-reported health-related quality-of-life instrument for people with multiple sclerosis. Subjects rate six quality-of-life domains: Mobility, Symptoms, Emotional well-being, General contentment, Thinking/fatigue, and Family/social well-being. Scores range from zero to 176; higher scores indicate better health-related quality of life. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include the FAMS scores acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed a baseline questionnaire were included.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 36 | 30 | 34
score on a scale | 0.056 [-0.277 to 0.389] | 0.051 [-0.357 to 0.459] | 0.240 [-0.087 to 0.567]

12. Other Pre Specified Outcome: Evaluation of How Overall Sleep Quality Impacts People With MS Using a Sleep Questionnaire (Pittsburgh Sleep Quality Index)
Description: The sleep questionnaire asks subjects to report various aspects related to their sleep routine. Scores range from zero to 21; higher score indicates worse sleep quality. In order to account for all contributed data (even for those who did not complete the study but contributed some post-randomization data in the active study phase), the analyses include the PSQIs acquired within the active treatment phase (from baseline to week 24 visit). We then calculated and report the average change per week in the score.
Time Frame: Up to week 24 visit
Population: Participants who completed the baseline assessment were eligible for inclusion.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
Number analyzed (Participants) | 34 | 30 | 33
score on a scale | -0.026 [-0.091 to 0.039] | 0.035 [-0.035 to 0.105] | -0.045 [-0.110 to 0.021]

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the point of randomization until a participant terminated from the study. Unresolved AEs, as well as SAEs, were followed for an added 30 days after study completion. Up to 48 weeks overall.
Description: Adverse events were captured through mixed methods. Subjects were provided with a diary in which to record adverse events. Serious adverse events that were catalogued as such due to hospital admission were also captured systematically if the admission occurred within our hospital system through automated reports to the PI. Other times, the adverse events were captured non-systematically, such as through ad hoc reports to study team members.
Arm/Group | Intranasal Insulin 20 International Units | Intranasal Insulin 10 International Units | Placebo
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 5/37 | 3/33 | 5/35
Other Adverse Events (participants affected / at risk) | 24/37 | 18/33 | 18/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intranasal Insulin 20 International Units (N=37) | Intranasal Insulin 10 International Units (N=33) | Placebo (N=35)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (2) | 1 (1)
Perirectal abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Non-epileptic seizure (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Worsening of neurological symptoms (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Zoster ophthalmicus (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Small bowel obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pain (Cardiac disorders) | 1 (5) | 0 (0) | 0 (0)
Multiple sclerosis relapse (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Intranasal Insulin 20 International Units (N=37) | Intranasal Insulin 10 International Units (N=33) | Placebo (N=35)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2
Fatigue (General disorders) | 1 | 2 | 1
Irritability (Psychiatric disorders) | 1 | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Headache (Nervous system disorders) | 8 | 5 | 5
Upper respiratory infection (Infections and infestations) | 1 | 3 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0 | 1
Nightmare (Psychiatric disorders) | 0 | 0 | 2
Pain (General disorders) | 2 | 1 | 4
Dizziness (Nervous system disorders) | 4 | 3 | 2
Fall (Injury, poisoning and procedural complications) | 2 | 1 | 1
Weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0
Memory impairment (Nervous system disorders) | 2 | 0 | 1
Fracture (Injury, poisoning and procedural complications) | 3 | 1 | 0
Paresthesia (Nervous system disorders) | 2 | 2 | 1
Diarrhea (Gastrointestinal disorders) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
This study faced major disruptions due to the COVID-19 pandemic. Per IRB, all in-person research activities were halted from mid-March until mid-July 2020. Remote study activities were conducted, where possible. 13 participants who were in the active treatment phase of the study stopped study drug early per DSMB. After re-opening, per IRB request, in-person study visits were restricted to the minimum needed for the main study goals. Thus, there is greater than anticipated missingness.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2020-11-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT02988401/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/01/NCT02988401/SAP_001.pdf
  • Informed Consent Form (2020-07-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT02988401/ICF_002.pdf